CLINICAL TRIAL: NCT05367817
Title: Effects of a Neuromuscular Joint Protective Exercise Therapy Program for Treatment of Wrist Osteoarthritis: a Randomized Controlled Trial
Brief Title: Effects of a Neuromuscular Exercise Therapy Program for Treatment of Wrist Osteoarthritis: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-02437; 2020-03807
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis Wrist
Keywords: Wrist Osteoarthritis, SLAC, SNAC, exercise therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy (Experimental): The program consists of two parts. The first part of the program contains unloaded active ROM exercises for the wrist in flexion/extension, radial-/ulnardeviation and pronation/supination. The second part of the program consists of three neuromuscular exercises that focus on coordination, wrist stability and strength. The participants will perform the program twice a day for 12 weeks.
  Interventions: Other: Neuromuscular exercise therapy
- Training program (Active Comparator): The training program for the control group will consist of ROM exercises only that will be also be performed twice a day for 12 weeks.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Neuromuscular exercise therapy — Participants perform specific neuromuscular exercises aimed at enhancing the sensorimotor control of the wrist.
  Arms: Exercise therapy
Other: Training program — Participants perform range of motion exercises for the wrist.
  Arms: Training program

SUMMARY:
Individuals with wrist osteoarthritis (OA) can suffer from pain, muscular weakness, and impaired motion of the wrist, which can reduce the quality of life. While there is strong evidence that all patients with OA should receive first-line treatment with education and exercises, this approach has not yet been proposed for individuals with wrist OA. Therefore, this trial aimed to evaluate the effectiveness of a first line neuromuscular joint protective exercise therapy program compared to a training program with range of motion (ROM) exercises in patients with wrist OA.

DETAILED DESCRIPTION:
Background: Post-traumatic wrist OA develops slowly, and the joint degeneration may eventually lead to pain, muscular weakness, and stiffness of the wrist. As a result, this can affect the function of the entire upper limb, which can interfere with activities of daily living and the ability to work; thus, leading to reduced quality of life. A progress of disproportionate joint load and disturbed neuromuscular control are frequently present and may even make the condition worse.

Exercise therapy has been defined as a regime of physical activities designed and prescribed for precise therapeutic goals, aiming at educating the performance of specific exercises to improve neuromuscular control, reduce pain and achieve functional joint stability.

Self-management programs, including exercise therapy and joint protective strategies, are core treatments in knee and hip OA. Since the complex wrist joint cannot fully be compared to larger weight-bearing joints as the knee and hip, there is a need to develop exercise therapy programs specially designed for the wrist. Such a program should be part of a comprehensive joint protective standard care and could be beneficial to decrease disability and postpone, or possibly even eliminate, the need for surgery in individuals with wrist OA.

Aim: This is a randomized controlled trial (RCT) with the aim to investigate if a self-managed exercise therapy program with joint protective strategies to improve neuromuscular control (intervention group) will reduce pain and improve function more compared to a training program with range of motion (ROM) exercises (control group).

Material and methods: This study is a single-blinded randomized controlled trial (RCT) in patients with symptomatic and radiographically verified wrist OA with two treatment arms. The participants will be randomly assigned either to an exercise therapy program (intervention group) or to a training program including ROM exercises only. The participants in both groups will receive structured education on 1) wrist anatomy; 2) pathophysiology; 3) joint protective self-management strategies and 4) management of pain and fatigue by exercises.

Both program will consist of home exercises twice a day for 12 weeks. The treatments will be followed up by the treating physiotherapist at the department of hand surgery in Malmö, Sweden at 2-, 6- and 12-weeks post baseline, and the participants will be contacted by telephone at 4 and 8 weeks post baseline. Assessments will be performed at baseline and at 3, 6, and 12 months after baseline by an independent assessor, who is blinded to the participants' group allocation. At the 3- and 6-months follow-up, the participants will rate their global rating of change (GROC) regarding how they perceive their wrist pre- and post-training.

ELIGIBILITY:
Inclusion criteria:

1. Radiographically confirmed and symptomatic wrist OA - SLAC and SNAC stage 1-3
2. Age≥18

Exclusion criteria:

1. The presence of other diseases or disorders that could affect arm and hand function
2. Previous surgery to the wrist
3. Intraarticular wrist cortisone injection within the last 3 months
4. Inability to understand and follow test instructions due to communicative, mental, or cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain and function on the Patient-Rated Wrist Evaluation (PRWE) at 3, 6 and 12 months. | Baseline, 3, 6 and 12 months
  The PRWE is a self-reported questionnaire that includes 15 questions, divided into two subscales assessing pain (5 items) and function (10 items, 6 concerning specific tasks and 4 the ability to perform daily activities) over the past week. The questions are scored on a 10-point ordered categorical scale, ranging from no pain or no difficulty (0 points), to worst pain or unable to do (10 points). The total score of the subscales pain (sum of 5 items) and function (sum of 10 items divided by 2) ranges from 0 to 50. The maximum total score of PRWE is 100 and represents the worst disability, whereas 0 represents no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Brogren, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsson SL, Ekstrand E, Dahlin LB, Bjorkman A, Brogren E. Effects of a neuromuscular joint-protective exercise therapy program for treatment of wrist osteoarthritis: a randomized controlled trial. BMC Musculoskelet Disord. 2024 Jan 5;25(1):38. doi: 10.1186/s12891-023-07157-4. PMID 38183045
- [Derived] Larsson SL, Ekstrand E, Dahlin LB, Bjorkman A, Brogren E. A self-managed exercise therapy program for wrist osteoarthritis: study protocol for a randomized controlled trial. Trials. 2023 Oct 2;24(1):628. doi: 10.1186/s13063-023-07668-4. PMID 37784197

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT05367817/Prot_SAP_000.pdf